CLINICAL TRIAL: NCT07170852
Title: Single Dose Oral Bioequivalence Study of Bempedoic Acid 180 mg Film Coated Tablet and Nilemdo® (Bempedoic Acid) 180 mg Film-coated Tablets in Healthy Adult Human Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Bempedoic Acid 180 mg Film Coated Tablet and Nilemdo® (Bempedoic Acid) 180 mg Film-coated Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Humanis Saglık Anonim Sirketi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: C1B05475
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Hypercholesterolaemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bempedoic acid film coated tablet (Experimental): Bempedoic acid 180 mg film coated tablet
  Interventions: Drug: Bempedoic acid film coated tablet; Drug: Nilemdo® Film-coated tablets
- Nilemdo® Film-coated tablets (Active Comparator): Nilemdo® (Bempedoic Acid) 180 mg Film-coated tablets
  Interventions: Drug: Bempedoic acid film coated tablet; Drug: Nilemdo® Film-coated tablets

INTERVENTIONS:
Drug: Bempedoic acid film coated tablet — 1 tablet of 180 mg Bempedoic Acid
Drug: Nilemdo® Film-coated tablets — 1 tablet of 180 mg Bempedoic Acid

SUMMARY:
Single dose oral bioequivalence study of Bempedoic Acid 180 mg Film Coated Tablet and Nilemdo® (Bempedoic Acid) 180 mg Film-coated tablets in healthy adult human subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 55 years old, both inclusive
* Sex: Males and/or non-pregnant, non-lactating females
* Female of childbearing potential had a negative serum beta human chorionic gonadotropin (β-HCG) pregnancy test performed within 28 days of the first dose of study medication. They used an acceptable form of contraception.

For female of childbearing potential, acceptable forms of contraception included the following:

* Non hormonal intrauterine device in place for at least 3 months prior to the start of the study and remaining in place during the study period, or
* Barrier methods containing or used in conjunction with a spermicidal agent, or
* Surgical sterilization, or
* Practicing sexual abstinence throughout the course of the study.
* Females were not considered of childbearing potential if one of the following was reported and documented on the medical history:
* Postmenopausal with spontaneous amenorrhea for at least one year, or
* Spontaneous amenorrhea for more than 6 months and less than one year with Serum Follicular Stimulating Hormone (FSH) level > 40 mIU/mL, or
* Bilateral oophorectomy with or without a hysterectomy and an absence of bleeding for at least 6 months, or
* Total hysterectomy and an absence of bleeding for at least 3 months.
* BMI: 18.5 to 30.0 kg/m2, both inclusive; BMI values were rounded off to one significant digit after decimal point (e.g. 30.04 rounds down to 30.0, while 18.45 rounds up to 18.5).
* Non-smokers and non-tobacco user (i.e. who had no past history of smoking and tobacco consuming for at least one year prior to study).
* Able to communicate effectively with study personnel.
* Able to give written informed consent to participate in the study.
* All volunteers were judged by the principal or sub-investigator or physician as normal and healthy during a pre-study safety assessment performed within 28 days of the first dose of study medication which included:
* A physical examination (clinical examination) with no clinically significant finding.
* Results within normal limits or clinically non-significant for the following tests

Exclusion Criteria:

* History of allergic responses to Bempedoic acid or other related drugs and any of its formulation ingredients.
* Had significant diseases or clinically significant abnormal findings during screening [medical history, physical examination (clinical examination), laboratory evaluations, ECG recording, gynecological history and examination (including pelvic examination and routine breast examination) (for female volunteers)].
* Any disease or condition like diabetes, psychosis or others, which might compromise the haemopoietic, gastrointestinal, renal, hepatic, cardiovascular, respiratory, central nervous system or any other body system.
* History or presence of bronchial asthma.
* Used any hormone replacement therapy within 3 months prior to the first dose of study medication.
* A depot injection or implant of any drug within 3 months prior to the first dose of study medication.
* Used CYP enzyme inhibitors or inducers within 30 days prior to the first dose of study medication (see https://druginteractions.medicine.iu.edu/MainTable.aspx).
* History or evidence of drug dependence or of alcoholism or of moderate alcohol use.
* History of difficulty with donating blood or difficulty in accessibility of veins.
* A positive hepatitis screen (includes subtypes B & C).
* A positive test result for HIV antibody.
* Subjects who had received a known investigational drug within seven elimination half-life of the administered drug prior to the first dose of study medication.
* Subject who had donated blood or loss of blood 50 ml to 100 ml within 30 days or 101 ml to 200 ml within 60 days or >200 ml within 90 days (excluding volume drawn at screening for this study) prior to first dose of study medication, whichever was greater.
* History of difficulty in swallowing or of any gastrointestinal disease, which could affect drug absorption.
* Intolerance to venipuncture.
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the principal investigator or sub-investigator, could contraindicate the volunteer's participation in this study.
* Institutionalized volunteer.
* Used any prescribed medications (including simvastatin and pravastatin) within 14 days prior to the first dose of study medication.
* Used any OTC products, vitamin and herbal products, etc., within 7 days prior to the first dose of study medication.
* Used of grapefruit and grapefruit containing products within 7 days prior to the first dose of study medication.
* Ingestion of any caffeine or xanthine products (i.e. coffee, tea, chocolate, and caffeine-containing sodas, colas, etc.), recreational drugs, alcohol or other alcohol containing products within 48 hours prior to the first dose of study medication.
* Ingestion of any unusual diet, for whatever reason (e.g.: low sodium) for three weeks prior to the first dose of study medication.
* Subject who had serum uric acid higher than the upper limit of normal range during screening.
* AST, ALT values are 1.1 times higher than the upper limit of normal range during screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2025-05-21 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2025-08-21 (Actual)

PRIMARY OUTCOMES:
Maximum measured plasma concentration (Cmax) | 72 hours
  To determine bioequivalence for bempedoic acid, the 90% confidence interval of the relative mean (geometric least squares mean) of the assay to the reference product for the Ln-transformed Pharmacokinetic parameters Cmax had to be between 80.00% and 125.00%.
Area under the plasma concentration versus time curve from the zero time point to the last quantifiable concentration (AUCt) | 72 hours
  The 90% confidence interval of the relative mean (Geometric least square mean) of test to reference product for Ln-transformed Pharmacokinetic parameters AUCt was to be within 80.00% to 125.00% for Bempedoic acid to establish bioequivalence.

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve from zero to infinity (AUCi) | 72 hours
  Descriptive Statistics
Time of the maximum measured plasma concentration (Tmax) | 72 hours
  Descriptive Statistics
Elimination Rate Constant (Kel) | 72 hours
  Descriptive Statistics
Apparent terminal elimination half-life (tHalf) | 72 hours
  Descriptive Statistics

CONTACTS AND LOCATIONS:
Locations (1):
- Cliantha Research Limited, Noida, India

IPD SHARING:
Plan to Share IPD: No